CLINICAL TRIAL: NCT06744309
Title: Heat Adaptation Through Community-based Approaches and Research at SEACO: Structural and Behavioural Interventions
Brief Title: Heat Adaptation Through Community-based Approaches and Research at SEACO: Structural and Behavioural Interventions (Heat Care)
Acronym: Heat Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University Malaysia (Other)
Collaborators: Monash University (Other); Heidelberg University (Other); Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Tin Tin Su, Professor, Monash University Malaysia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: MUHREC43232
Record Dates: First submitted 2024-12-11; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Climate Change; Heat; Weather; Heat Effect; Heat; Excess
Keywords: heat health; heat literacy; thermotolerance; Rising average temperature
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: The study uses a 2 x 2 factorial design to evaluate the effectiveness of cool roofs and heat literacy education in mitigating extreme heat impacts in rural Malaysian communities. Participants, randomly selected from the SEACO database, will be divided into four groups: both interventions, cool roof only, heat literacy only, and control. Cool roofs involve painting roofs with UV-resistant white paint to reduce heat absorption, while heat literacy includes 8-12 weeks of education on heat awareness and personal cooling strategies. Data will be collected at baseline, 3, 6, and 12 months through surveys, physical measurements, and Garmin Vivosmart 5 wearable sensor and SwitchBot meter. The primary endpoints are indoor temperature, physical activity (step count), glycemic control (HbA1c) and sleep duration. The study aims to develop an evidence-based, culturally sensitive community heat adaptation program to improve heat resilience in rural Malaysia.
Masking Description: No, the study does not involve masking (blinding). Due to the nature of the interventions-cool roof installation and heat literacy education-it is not possible to blind the participants or the field team members (including researchers). However, the random selection and assignment of participants to intervention and control groups will be conducted by a statistician who is not part of the research team, ensuring an unbiased allocation process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Cool Roof and Heat Literacy Interventions) (Active Comparator): Cool roof intervention: Roofs will be painted with UV-resistant paint to reduce thermal absorption.
  Heat literacy intervention: Participants will receive education and training on heat-related health risks and coping strategies.
  Interventions: Behavioral: Heat Literacy Intervention; Other: Structural (Cool Roof) Intervention
- Group B (Cool Roof Intervention Only) (Active Comparator): Cool Roof intervention: Roofs will be painted with UV-resistant white paint to reduce thermal absorption
  Interventions: Other: Structural (Cool Roof) Intervention
- Group C (Heat Literacy Intervention Only) (Active Comparator): -Heat literacy intervention: Participants will receive education and training on heat-related health risks and coping strategies.
  Interventions: Behavioral: Heat Literacy Intervention
- Group D (Control Group) (No Intervention): No intervention will be provided, serving as a control group for comparison.

INTERVENTIONS:
Behavioral: Heat Literacy Intervention — The behavioral intervention aims to improve heat literacy among participants through an 8-12 week education and training program. It includes three main modules: enhancing community awareness of hot weather, recognizing and responding to heat-related illnesses, and teaching personal cooling strategies. Participants will use SwitchBot meters to monitor indoor temperature and humidity, access real-time weather information, and learn about heat wave warnings. They will receive educational materials, including infographics, videos, and one-to-one training from field staff. The content of intervention and delivery methods will be refined through co-design workshops with stakeholders and community members to ensure they are practical and culturally appropriate. The goal is to equip participants with the knowledge and skills to protect themselves from extreme heat, resulting in better heat adaptation behaviors and improved health outcomes.
  Arms: Group A (Cool Roof and Heat Literacy Interventions); Group C (Heat Literacy Intervention Only)
Other: Structural (Cool Roof) Intervention — The structural intervention in this study involves implementing cool roofs to reduce indoor temperature and mitigate the effects of extreme heat in rural Malaysian communities. Selected households will have their roofs painted with UV-resistant paint, which reflects direct sunlight and reduces thermal absorption. This intervention aims to decrease the amount of solar energy absorbed by the roof, thereby lowering indoor temperature and reducing the physiological heat strain on residents. By maintaining cooler indoor environment, the cool roof intervention seeks to alleviate the health risks associated with prolonged exposure to high temperature.
  Arms: Group A (Cool Roof and Heat Literacy Interventions); Group B (Cool Roof Intervention Only)

SUMMARY:
The goal of this clinical trial is to learn if structural and behavioral interventions can mitigate the health effects of extreme heat in rural Malaysian communities. The study focuses on implementing cool roofs (a passive cooling system) and heat literacy education to improve heat adaptation behaviors. The main questions it aims to answer are:

* Does the implementation of cool roofs reduce indoor temperatures and related heat stress in rural households?
* Does heat literacy education improve community awareness and behaviors related to coping with extreme heat?

Researchers will compare four groups: one receiving both cool roofs and heat literacy interventions, one receiving only the cool roof intervention, one receiving only heat literacy education, and a control group receiving neither intervention. Participants will be asked to:

* Have their roofs painted with UV-resistant white paint (for cool roof intervention groups).
* Participate in educational sessions and training on heat-related health risks and coping strategies (for heat literacy intervention groups).
* Complete baseline and follow-up surveys at 3, 6, and 12 months.
* Wear a Garmin Vivosmart 5 sensor for two weeks during each data collection period to monitor heart rate, physical activity, and sleep patterns.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the effectiveness of structural and behavioral interventions in mitigating the health impacts of extreme heat in rural Malaysian communities. Specifically, the study will implement and assess two interventions: cool roofs (a passive cooling system) and heat literacy education. Cool roofs involve painting the roofs of selected households with UV-resistant white paint to reduce thermal absorption, thereby lowering indoor temperatures. Heat literacy education aims to enhance community awareness and preparedness for extreme heat by providing training and educational materials on recognizing heat-related illnesses and adopting personal cooling strategies.

Participants will be randomly selected from the SEACO health database, encompassing five operational sub-districts. Eligible participants include adults aged 18 years and above, living in single-story houses with suitable roofing materials. They will be randomly assigned to one of four groups: one receiving both interventions, one receiving only the cool roof intervention, one receiving only heat literacy education, and a control group receiving neither intervention. This 2 x 2 factorial design will allow researchers to compare the effects of each intervention individually and in combination.

Data collection will occur at baseline and three follow ups, intended to do 3 months, 6 months, and 12 months. SEACO data collectors will visit participants' homes to install SwitchBot heat and humidity measurement devices, conduct surveys, and take physical measurements. Participants will also wear Garmin Vivosmart 5 sensors for two weeks during each data collection period to monitor their heart rate, physical activity, and sleep patterns. We will also conduct the basic measurements such as height, weight, blood pressure, blood glucose and HbA1c. The surveys will gather information on socioeconomic and demographic characteristics, self-reported illnesses, heat exposure, heat adaptation behaviors, heat literacy, cooling strategies, self- reported sleep quality, mental health and quality of life.

The study aims to determine whether cool roofs and heat literacy education can effectively reduce indoor temperatures, improve heat adaptation behaviors, and ultimately mitigate the health risks associated with extreme heat. By analyzing data from both interventions and their combined effect, the research seeks to develop a theoretically informed, evidence-based, and culturally sensitive community-based heat adaptation program for rural Malaysia. This program could serve as a model for other climate-vulnerable regions, providing valuable insights into sustainable and practical approaches to addressing the health impacts of climate change.

ELIGIBILITY:
Individual Inclusion Criteria:

* Adults aged at least 18 years old
* Willing to participate in all study components
* Consent to roof painting and installation of heat and humidity measurement devices
* Consent to wear the supplied wearables (Garmin Vivosmart 5) for data collection
* No plans to relocate during the study period
* Possess a smartphone for receiving health education materials

Individual Exclusion Criteria:

* Individuals belonging to one household with existing participants
* Bedridden individuals or those requiring assistance in movement

Household Inclusion Criteria:

* Single-story house
* Main house measurement less than 1200 sqft
* Built with brick or brick and wooden
* Roof made of zinc, ceramic/clay, or mixed, suitable for cool roof painting
* Minimal to no requirement for roof repair
* No plans for renovation during the study period

Household Exclusion Criteria:

* Double-story houses, shops, or empty houses
* Houses with the facility to sprinkle water on the roof

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Indoor Air Temperature | 12 months
  Assessed using an indoor data logger (SwitchBot) to measure air temperature within the household.
Step count (Physical Activity) | 12 months
  Tracked using Garmin Vivosmart 5 sensors, recording steps and distance.
Sleep Duration | 12 months
  This will be obtained using the Uppsala Sleep Inventory questionnaire which assess sleep duration.
Glycaemic Control | 12 months
  HbA1c level which will be measured by the Hemocue® HbA1c 501 System.

SECONDARY OUTCOMES:
Depressive Symptoms | 12 months
  This will be assessed using the Quick Inventory of Depressive Symptomatology (QIDS-SR16) questionnaire.
  The Quick Inventory of Depressive Symptomatology (QIDS-SR16) assesses the severity of depressive symptoms based on 16 items. The scoring for the QIDS-SR16 is as follows:
  Minimum possible score: 0 Maximum possible score: 27
  A higher score on the QIDS-SR16 indicates more severe depressive symptoms, which means a worse outcome in terms of depression severity. Conversely, lower scores suggest fewer symptoms and thus a better outcome.
Psychological Distress | 12 months
  This will be assessed using the Kessler Psychological Distress Scale (K10) questionnaire.
  The Kessler Psychological Distress Scale (K10) is a tool used to measure psychological distress. It consists of 10 items, each rated on a 5-point scale from "none of the time" (score = 1) to "all of the time" (score = 5).
  Minimum possible score: 10 (if the participant scores "none of the time" for all 10 items).
  Maximum possible score: 50 (if the participant scores "all of the time" for all 10 items).
  Higher scores on the K10 indicate greater psychological distress (worse outcomes)
Heat-related Illnesses | 12 months
  This outcome tracks the incidence and severity of heat-related illnesses among participants, such as heat exhaustion and heat stroke. Data is collected through self-reported health metrics. The goal is to identify any reductions in heat-related illnesses due to the interventions.
Health-related Quality of Life | 12 months
  This outcome evaluates the overall well-being of participants using the EuroQol five dimensions of health (EQ-5D) questionnaire, which covers five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The assessment aims to determine how the interventions impact participants' overall quality of life and well-being. The minimum value is 0 and maximum value is 100.
  Higher scores generally indicate better health outcomes, meaning that the person is in a state of better physical and mental health.
  Lower scores indicate worse health outcomes or greater health problems.
Indoor Thermal Comfort | 12 months
  Assessed using a visual analogue scale to measure current heat experience in the household rated on a visual scale from: Very comfortable, Comfortable, Just comfortable, Just uncomfortable, Uncomfortable, and Very uncomfortable. Minimum (1) to maximum (6). The higher score is the worse outcome.
Heat Adaptation Practices | 12 months
  This outcome evaluates participants' adaptive behaviors during periods of extreme heat, highlighting measures taken to protect themselves and their communities from heat-related health impacts. The 18-item questionnaire evaluates heat adaptation practices using a 5-point Likert scale (1 = Strongly Disagree to 5 = Strongly Agree). Negatively worded statements will be reversed. Scores range from 18 to 90, with higher scores indicating higher adoption in heat adaptation practices, and lower scores indicating lower adoption in heat adaptation practices.

OTHER OUTCOMES:
Heat Index | 12 months
  Assessed using an indoor data logger (SwitchBot) to measure heat index within the household.
Blood Glucose Level | 12 months
  Random blood glucose, which will be measured using a home blood glucose monitoring system (Accu Chek Instant S)
Sleep Inventory | 12 months
  This will be obtained using the Uppsala Sleep Inventory questionnaire, which assesses an individual's difficulty initiating sleep, maintaining sleep, and individual's daytime sleepiness.
Heat Literacy | 12 months
  This outcome assesses participants' ability to access, understand, appraise, and apply information to make judgments and take decisions in everyday life to mitigate heat effects on health using structured questionnaire. The index is standardized to unified metrics from 0 to 50. 0 represents the lowest heat literacy and 50 the highest heat literacy.

CONTACTS AND LOCATIONS:
Overall Officials: Tin Tin Su, MBBS, Dr.Med, Principal Investigator — Monash University Malaysia
Locations (1):
- South East Asia Community Observatory, Monash University Malaysia, Segamat, Johor, Malaysia

IPD SHARING:
Plan to Share IPD: No
No There is no plan to make IPD available. The MUHREC requirement to comply with the term "Retention and storage of data - The Chief Investigator is responsible for the storage and retention of the original data pertaining to the project for a minimum period of five years".